CLINICAL TRIAL: NCT02710565
Title: Use of Endo Bronchial Ultrasound (EBUS) Trans Bronchial Needle Aspiration (TBNA) for Cell Culture as an Aid to Diagnose Lung Cancer and Lymphoma
Brief Title: Use of EBUS TBNA for Cell Culture as an Aid to Diagnose Lung Cancer and Lymphoma
Acronym: EBUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B723
Record Dates: First submitted 2016-03-07; First posted 2016-03-17 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Lung Cancer; Lymphoma; Non-small Cell Lung Cancer; Non-Hodgkin Lymphoma; Mediastinal Lymphadenopathy
Keywords: Endo bronchial ultrasound; Trans bronchial needle aspiration; Cell line; Lung cancer
MeSH Terms: conditions — Lung Neoplasms; Lymphoma; Carcinoma, Non-Small-Cell Lung; Lymphoma, Non-Hodgkin | interventions — Cohort Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort (Other): Participants who are scheduled to have an endo bronchial ultrasound (EBUS) trans bronchial needle aspiration (TBNA) will provide additional samples. These samples will then be sent to Imperial College London to see whether a cell line can be grown.
  If growth is successful then the samples will be returned to our pathology department to see if grading is possible and then to compare these results with the previous diagnostic samples.
  The cell line samples will not be used for patient diagnosis.
  Interventions: Other: Cohort

INTERVENTIONS:
Other: Cohort — Obtaining additional EBUS TBNA samples for cell culture
  Other Names: EBUS TBNA

SUMMARY:
Participants who are scheduled to have an endo bronchial ultrasound (EBUS) trans bronchial needle aspiration (TBNA) will provide additional samples. These samples will then be sent to Imperial College London to see whether a cell line can be grown.

If growth is successful then the samples will be returned to our pathology department to see if grading is possible and then to compare these results with the previous diagnostic samples.

The cell line samples will not be used for patient diagnosis.

DETAILED DESCRIPTION:
Obtaining adequate pathological specimen is essential in the diagnosis of cancer. Ultrasound guided sampling through endo bronchial ultrasound (EBUS) trans bronchial needle aspiration (TBNA) has emerged as a safe and accurate technique in the diagnosis and staging of lung cancer but subtyping and/or genotyping of TBNA samples obtained by convex probe EBUS has long been considered to be limited by the lack of tissue architecture in these small tissue samples. The performance of small tissue samples in non-small cell lung cancer (NSCLC) subtyping has been proven to be accurate in modern pathology practice adopting cell blocks and immunohistochemistry (IHC), reducing the NSCLC not otherwise specified rate for needle aspiration samples to 8-23%. It has also shown recently a promising result in work up of mediastinal lymphadenopathy when lymphoma is suspected.

It is thought that at times EBUS TBNA sample is still inadequate for further essential testing for diagnostic and therapeutic purpose and enhancing the yield is possibly by cell culture will not only be useful for diagnosing lung cancer and lymphoma but also will provide material for future research study.

We have therefore developed a research proposal in collaboration with scientists at the biomedical research laboratory at Imperial College London, who have excellent record in basic scientific research and currently involved in similar research on cell culture for other type of diseases.

ELIGIBILITY:
Inclusion criteria

1. Male or females aged >18 years
2. Completed Chest CT
3. Written informed consent

Exclusion criteria

1. Patients with active tuberculosis (TB)
2. Pregnancy
3. Patients with significant psychiatric and or neurological comorbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-02; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Cell culture growth | upto 50 Weeks
  Are samples from EBUS TBNA suitable for cell culture?

SECONDARY OUTCOMES:
Diagnostic benefit | upto 50 Weeks
  To ascertain the diagnostic benefit of EBUS TBNS for diagnosis of lymphoma in patients with isolated mediastinal lymphadenopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Dipak Mukherjee, MRCP MBBS, Principal Investigator — Mid and South Essex NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Basildon Hospital, Basildon, Essex
  - Imperial College London, London

IPD SHARING:
Plan to Share IPD: No